CLINICAL TRIAL: NCT06525844
Title: Clinical and Radiographic Outcomes With the Use of I-PRF in Mature Permanent Teeth With Symptomatic Irreversible Pulpitis : A Randomized Control Trial
Brief Title: Regenerative Endodontic Therapy in Cases of Irreversible Pulpitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Shahbaz Saqib, Doctor, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSaqib
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Symptomatic Irreversible Pulpitis
MeSH Terms: interventions — Blood Coagulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- regenerative endodontic therapy with blood clot (Active Comparator): In the procedures of regenerative endodontics therapy, K-files were intentionally used to violate the periapical tissues via overinstrumentation up to 2-3mm past the apical foramen to induce bleeding. The adequate blood need to be full with canal space and below the CEJ, then wait for 10-15min to coagulate.
  Interventions: Procedure: blood clot
- regenerative endodontic therapy with I-PRF (Experimental): In the procedures of regenerative endodontics therapy, K-files were intentionally used to violate the periapical tissues via overinstrumentation up to 2-3mm past the apical foramen to induce bleeding. Only the apex 1/3 of the root canal need to be filled with blood. PRF was injected into the root canal to a level below the CEJ, then wait for 10-15min to coagulate.
  Interventions: Procedure: regenerative endodontic therapy using I-PRF

INTERVENTIONS:
Procedure: regenerative endodontic therapy using I-PRF — Blood will be taken from medial cubital vein
  Arms: regenerative endodontic therapy with I-PRF
Procedure: blood clot — Other: BC According to the procedures of regenerative endodontics therapy, BC was made by the way of provoking apical bleeding into root canal.
  Arms: regenerative endodontic therapy with blood clot

SUMMARY:
Root canal therapy (RCT) is a classical and effective treatment that is currently utilised in dental practice, offering high success rates for pulp and periapical diseases; however, teeth after RCT are susceptible to altered pulp defence and sensory function, even fractures, as a consequence of pulp loss. Furthermore, several studies have highlighted that the actual failure rate of standard root canal treatments performed in general practice is significantly higher than expected . Moreover, these treatments are lengthy and costly and are often subject to retreatment .Inherent in this procedure(rct) is loss of dental hard tissue and subsequent weakening of the treated tooth,making them more prone to fracture. Therefore, less invasive alternative strategies could be used to treat pulpitis, even when irreversible.

Murray et al. proposed the term "Regenerative endodontic treatment (RET)" in 2007, based on a tissue engineering concept (stem cells, biomimetic scaffolds, and bioactive growth factors). The 2016 American Association of Endodontists (AAE) guidelines formally defined RET as a collection of "biologically based procedures designed to replace damaged tooth structures, including dentine and root structures, as well as cells of the pulp-dentine complex"

DETAILED DESCRIPTION:
Mature permanent teeth with Irreversible Pulpitis have traditionally been managed with root canal treatment .However this procedure significantly reduces the survival rate of tooth. Acknowledging the inherent healing potential of an infection-free pulp, attempts have been made to use pulpotomy as a treatment modality in permanent teeth with complete root development exhibiting symptoms of irreversible pulpitis, where the radicular pulp is still healthy. Besides, the issues associated with coronal pulpotomy in permanent teeth are uncertainty on the pulpal status at the time of treatment, and lack of predictability. Moreover, there is a dearth of information in the literature that assesses the healing potential of pulp tissue in terms of clinical and radiographic outcomes in mature teeth with irreversible pulpitis.Regenerative endodontic therapy (RET) has attracted increasing attention with the development of tissue engineering. RET applies the concept of tissue engineering to achieve revascularization, innervation, and restoration of odontoblastic layers. Unlike root canal therapy, the disinfected canals are filled with vital tissue in RET rather than biocompatible, nonvital foreign materials. While several studies have explored the potential of pulp regeneration for infected teeth, most studies are limited to the treatment of immature necrotic teeth . For mature permanent teeth, the vital pulp is also of great importance in enhancing the immune system in root canals, promoting dentin deposition under chronic stimuli, and preventing discolouration. However, most of the reports of pulp regeneration in mature teeth are case reports or case series as mature teeth have fewer stem/progenitor cells, have narrower apical pathways for cell migration, and are more difficult to disinfect. Hence, it is of great urgency to develop an improved RET procedure to maximise the regeneration potential of mature teeth and extend the indications of RET.

ELIGIBILITY:
Inclusion Criteria:

* Patients from both genders with an age range of 18-35 years old.
* Permanent teeth with mature roots with a diagnosis of irreversible pulpitis, with absorption damage to the apex, and the diameter of the apical hole is greater than 1 mm.
* A restorable tooth.
* There is no need to leave space for the final post/core restoration.
* Anterior teeth and premolars with single canal.
* A cooperative and compliant patient.
* Patients not allergic to the drugs and antibiotics which needed to complete treatment.
* No periodontal disease or root cracking.

Exclusion Criteria:

* Patients with other serious organ diseases, such as cardiopulmonary, kidney and other major diseases.
* Pregnant women or lactating or expecting within a year.
* Patients with apical cysts.
* Patients with poor cooperation and those who quit the study halfway.
* Patients with periodontitis.
* Patients with dental dysplasia or other oral genetic disorders.
* Patients with dental phobia.
* Patients with mental disorders.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Success of regenerative endodontics therapy | 12 months
  Success: Defined as clinical and radiographic assessment of the teeth. Clinical examination showed absence of clinical signs of pain and soft tissue pathology (e.g. abscess, sinus tract etc.). Radiographic assessment showed the reduction and/or absence of periapical radiolucency.

SECONDARY OUTCOMES:
Change in pulp vitality | 1、3、6、12 months
  Change in pulpal vitality will be assessed through pulpal response to sensitivity tests (cold, hot and electrical test) in teeth treated with RET.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shahbaz Saqib, BDS, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University
Locations (1):
- Dr Shahbaz Saqib, Islamabad, ICT, Pakistan

IPD SHARING:
Plan to Share IPD: No